CLINICAL TRIAL: NCT07199036
Title: Clinical Application of the Effect of Respiratory Muscles Electrical Stimulation on Weaning in Patients With Difficult Weaning of the Mechanical Ventilation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Collaborators: Beijing Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Yi Li, Principal Investigator, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025bkky
Record Dates: First submitted 2025-09-29; First posted 2025-09-30 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Mechanical Ventilation
Keywords: Prolonged Mechanical Ventilation; transcutaneous phrenic nerve electrical stimulation; abdominal functional electrical stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (Sham Comparator): Sham TEDS + Sham abFES + Standard Care
  Interventions: Device: Sham TEDS; Device: Sham abFES
- TEDS Only (Experimental): TEDS + Sham abFES
  Interventions: Device: TEDS (Transcutaneous Diaphragmatic/Phrenic Nerve Stimulation); Device: Sham abFES
- abFES Only (Experimental): abFES + Sham TEDS
  Interventions: Device: abFES (Functional Electrical Stimulation of Abdominal Muscles); Device: Sham TEDS
- Combined (Experimental): TEDS + abFES
  Interventions: Device: TEDS (Transcutaneous Diaphragmatic/Phrenic Nerve Stimulation); Device: abFES (Functional Electrical Stimulation of Abdominal Muscles)

INTERVENTIONS:
Device: TEDS (Transcutaneous Diaphragmatic/Phrenic Nerve Stimulation) — Per session 20 min, twice daily; 5 days/week; up to 28 days or until successful weaning.
  Arms: Combined; TEDS Only
Device: abFES (Functional Electrical Stimulation of Abdominal Muscles) — Per session 20 min, twice daily
  Arms: Combined; abFES Only
Device: Sham TEDS — Position/time matched; 2 Hz low-intensity sensation only; no visible contraction.
  Arms: Control; abFES Only
Device: Sham abFES — Position/time matched; sensation only; no visible contraction.
  Arms: Control; TEDS Only

SUMMARY:
This trial evaluates whether transcutaneous diaphragmatic/phrenic nerve stimulation (TEDS), abdominal functional electrical stimulation (abFES), or their combination, accelerates and improves the quality of weaning from prolonged invasive mechanical ventilation (IMV), compared with standardized ICU care with sham stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Invasive mechanical ventilation ≥21 days for PMV; expected ≥48 h ICU stay. Eligible for standardized weaning protocol and SBT assessment. Informed consent by participant or legally authorized representative.

Exclusion Criteria:

* Non-screenable/unstable arrhythmia or hemodynamics; refractory hypoxemia/hypercapnia.

Pacemaker/ICD not shieldable; seizure disorder uncontrolled. Recent abdominal surgery or skin breakdown at electrode sites; BMI>35; pregnancy.

Prone positioning; continuous deep neuromuscular blockade; investigator deems unsuitable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-09-29 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Time to Successful Weaning (days) | From randomization up to Day 28
  Days from randomization to first day achieving ≥48 h free from invasive mechanical ventilation (IMV).

SECONDARY OUTCOMES:
Change in Diaphragm Excursion (DE) Measured by M-mode Ultrasound from Baseline to Day 28 (cm) | Baseline (within 24 hours before randomization) and Day 28 after randomization
  Diaphragm excursion will be measured by M-mode ultrasonography on the right hemidiaphragm. A 3.5-5.0 MHz convex probe is placed in the right subcostal region between the mid-clavicular and anterior axillary lines. The excursion (cm) during spontaneous breathe will be recorded as the average of three consecutive breaths. The outcome is the change in excursion from baseline to Day 28.
Change in Diaphragm Thickening Fraction (TFdi) from Baseline to Day 28 (%) | Baseline to Day 28
  Diaphragm thickness will be measured in the zone of apposition of the right hemidiaphragm with a high-frequency linear probe in B-mode. Thickness at end-expiration and end-inspiration will be recorded as the average of three breaths. The diaphragm thickening fraction (TFdi, %) is calculated as: (Thickness at end-inspiration - Thickness at end-expiration) / Thickness at end-expiration × 100. The outcome is the change in TFdi from baseline to Day 28.
Change in Diaphragm Thickness (DT) Measured by B-mode Ultrasound from Baseline to Day 28 (mm) | Baseline to Day 28
  Diaphragm thickness (mm) will be measured in the zone of apposition of the right hemidiaphragm using a high-frequency linear probe (7-12 MHz) in B-mode at end-expiration. The value is the average of three consecutive breaths. The outcome is the change in diaphragm thickness from baseline to Day 28.
Weaning Success From Invasive Mechanical Ventilation Within 28 Days (% of Participants) | Up to Day 28 after randomization
  Weaning success is defined as remaining free from invasive mechanical ventilation for at least 48 hours after extubation or tracheostomy decannulation. The outcome is the proportion of randomized participants who achieve successful weaning within 28 days after randomization.
28-Day In-hospital Cost From Randomization (CNY) | exactly 28 days
  Total in-hospital cost (Chinese Yuan) during the first 28 days after randomization
Change in PEF from Baseline to Day 28 (L/min) | Baseline to Day 28
Readmission | Readmission of 3 month/6 month/ 12 month
mortality | mortality of 3 month/6 month/ 12 month
Incidence of pulmonary infection | Incidence of pulmonary infection of 3 months/ 6 months/ 12 months
Ventilator-Free Days to Day 28 (VFDs-28) | Day 0-28 after randomization

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Rehabilitation Hospital, Capital Medical University, Beijing, Shijingshan District, China

IPD SHARING:
Plan to Share IPD: No